CLINICAL TRIAL: NCT05362747
Title: ProduceRx: Improving Weight and Cardiovascular Risk in Adults With Food Insecurity and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 851009
Record Dates: First submitted 2022-04-26; First posted 2022-05-05 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Obesity
Keywords: food insecurity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProduceRx (Experimental): Participants in the ProduceRx intervention group will be provided with BWL and produce vouchers for fresh fruits and vegetables.
  Interventions: Behavioral: Behavioral weight loss and produce vouchers
- Waitlist Control (No Intervention): Participants in the WLC group with be asked to stay weight stable, not to make changes in their eating and physical activity behaviors, and not to seek treatment for weight or eating during the waiting period.

INTERVENTIONS:
Behavioral: Behavioral weight loss and produce vouchers — Participants will receive weekly 30-minute, individual, in-person lifestyle counseling delivered by trained interventionists (e.g., registered dietitians) that consists of behavioral, dietary, and physical activity counseling. ProduceRx vouchers will be in the form of Food Bucks and will be provided at each session.
  Arms: ProduceRx

SUMMARY:
This is a pilot randomized controlled trial to assess the effects of providing produce vouchers during behavioral weight loss treatment in 40 adults with obesity and food insecurity. Participants will be randomized to ProduceRx (12 weekly sessions of in-person, behavioral weight loss counseling (BWL) + produce prescriptions) or a waitlist control (WLC).

DETAILED DESCRIPTION:
The proposed investigation is a single-site, pilot RCT to assess the effect of BWL and produce vouchers (ProduceRx) on diet quality, weight loss and cardiovascular risk factors among adult participants with food insecurity and obesity. Adults (N=40) will be randomized to a 12-week program that provides weekly, 30-minute BWL sessions + produce vouchers (n=20) or WLC (n=20). Outcomes will be assessed at baseline and at 12 weeks and include questionnaires, and measurements of weight, height, and cardiometabolic risk factors (blood pressure, waist circumference, and pulse). Participants will also be asked to complete two 24-hour dietary recalls.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. BMI ≥ 30 kg/m2
3. Food insecurity as assessed by the two-item "hunger vital sign"
4. Subjects must:

   1. have reliable telephone or Internet service to communicate with study staff
   2. plan to remain in the Philadelphia area for the next 6 months or more
5. Understand and be willing to comply with all study-related procedures and agree to participate in the study by giving written informed consent.

Exclusion Criteria:

1. Pregnant, nursing, or plans to become pregnant in the next 6 months
2. Serious medical risk such as uncontrolled diabetes, cancer, congestive heart failure, or recent cardiac event (e.g., myocardial infarction or stroke within the past 6 months)
3. Clinically significant hepatic or renal disease
4. History of (or plans for) bariatric surgery
5. Current psychiatric disorder that significantly interferes with daily living
6. Self-reported alcohol or substance abuse within the past 12 months
7. Use in past 3 months of medications known to induce significant weight loss (i.e., prescription weight loss medications) or weight gain (e.g., chronic use of oral steroids, second generation antipsychotics)
8. Loss of ≥ 10 lb of body weight within the past 3 months
9. Participation in a structured weight loss program in the prior 6 months
10. Inability to walk 2 blocks comfortably or engage in some other form of aerobic activity (e.g., swimming)
11. Participant from same household
12. Inability to attend treatment and/or assessment visits
13. Lack of capacity to provide informed consent
14. Any serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the patient's safety or successful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Dietary quality | Baseline, 12 weeks
  Change from baseline to 12 weeks in dietary quality from 24-hour dietary recalls summarized into Healthy Eating Index (HEI) Scores and caloric intake. Scores range from 0 to 100 with higher scores indicating better diet quality.

SECONDARY OUTCOMES:
Percent initial weight loss | Baseline, 12 weeks
  Change from baseline to 12 weeks in percent initial weight loss
Systolic blood pressure | Baseline, 12 weeks
  Change from baseline to 12 weeks in systolic blood pressure
Diastolic blood pressure | Baseline, 12 weeks
  Change from baseline to 12 weeks in diastolic blood pressure
Waist circumference | Baseline, 12 weeks
  Change from baseline to 12 weeks in waist circumference
Pulse | Baseline, 12 weeks
  Change from baseline to 12 weeks in pulse rate
Health-related quality of life | Baseline, 12 weeks
  Change from baseline to 12 weeks in general health-related quality of life (Short-Form-36). Scores range from 0 to 100 with higher scores indicating better quality of life.
Weight-related quality of life | Baseline, 12 weeks
  Change from baseline to 12 weeks in weight-related QOL (Impact of Weight on Quality of Life-Lite). Scores range from 0 to 100 with higher scores indicating better quality of life.
Food security | Baseline, 12 weeks
  Change from baseline to 12 weeks in the USDA Food Security Survey. Scores range from 0-10 with higher scores indicating lower food security.
Depressive symptoms | Baseline, 12 weeks
  Change from baseline to 12 weeks in Patient Health Questionnaire-8 Scores. Scores range from 0 to 24 with higher scores indicating more depressive symptoms.
Food addiction | Baseline, 12 weeks
  Change from baseline to 12 weeks in Yale Food Addiction Scores. Symptom scores range from 0 to 11 with higher scores indicating more symptoms.
Eating behaviors | Baseline, 12 weeks
  Change from baseline to 12 weeks in Eating Behaviors. Higher scores indicate greater agreement.
Self-regulation of eating | Baseline, 12 weeks
  Change from baseline to 12 weeks in self-regulation of eating as measured by the Regulation of Eating Behavior Scale. Scores range from 24 to 168 with higher scores indicating more self-regulation.
Self-regulation of exercise | Baseline, 12 weeks
  Change from baseline to 12 weeks in Behavioral Regulation in Exercise Questionnaire. Scores range from 0 to 76 with higher scores indicating more self-regulation.
Self-efficacy | Baseline, 12 weeks
  Change from baseline to 12 weeks in scores on the Weight Efficacy Lifestyle Questionnaire. Total scores range from 0 to 180. Higher scores represent greater eating self-efficacy.
Physical activity | Baseline, 12 weeks
  Change from baseline to 12 weeks in scores on the International Physical Activity Questionnaire. Higher scores indicate more physical activity.
Perceived Stress Scale | Baseline, 12 weeks
  Change from baseline to 12 weeks in scores on the Perceived Stress Scale. Scores range from 0-56 with higher scores indicating more stress.

CONTACTS AND LOCATIONS:
Overall Officials: Ariana M Chao, PhD, CRNP, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No